CLINICAL TRIAL: NCT02750748
Title: Pharmacokinetic Evaluation of Intranasal, Intramuscular, and Oral Naltrexone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Naltexone-Ph1a-002
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 4mg Intranasal Naltrexone (Experimental): Administer one 0.1 mL spray of a 40 mg/mL solution in one nostril
  Interventions: Drug: Naltrexone
- 4mg Intranasal Naltrexone with Intravail (Experimental): Administer 0.1 mL spray of a 40 mg/mL solution with 0.25% Intravail in one nostril
  Interventions: Drug: Naltrexone; Other: Intravail
- 2mg Intramuscular Naltrexone (Experimental): Administer 2 mg formulation intramuscularly
  Interventions: Drug: Naltrexone
- 50mg Naltrexone (Experimental): Administer 50mg formulation orally
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone
Other: Intravail
  Arms: 4mg Intranasal Naltrexone with Intravail

SUMMARY:
To determine the pharmacokinetics of 2 intranasal doses and 1 oral dose of naltrexone compared to an intramuscular dose of naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 55 years of age, inclusive.
* Provide written informed consent.
* BMI ranging from 18 to 30 kg/m2, inclusive.
* Adequate venous access.
* No clinically significant concurrent medical conditions determined by medical history, physical examination, clinical laboratory examination, vital signs, and 12-lead ECG.
* Male subjects must agree to use an acceptable method of contraception with female partners as well as not to donate sperm throughout the study and for 90 days after the last study drug administration. Female subject of childbearing potential must agree to use an acceptable method of birth control throughout the study and for 30 days after the last study drug administration. Oral contraceptives are prohibited.
* Agree not to ingest alcohol, drinks containing xanthine >500 mg/day (e.g., Coca Cola®, coffee, tea, etc.), or grapefruit/grapefruit juice.
* Participate in strenuous exercise 72 hours prior to admission through the last blood draw of the study.

Exclusion Criteria:

* Please contact site for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration (Cmax) | 48 hours
  Measurement of serum naltrexone prior to dosing and at times 2, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 hours after naltrexone administration
Plasma Concentration (Tmax) | 48 hours
  Measurement of serum naltrexone prior to dosing and at times 2, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 hours after naltrexone administration
Plasma Concentration (AUC 0-t) | 48 hours
  Measurement of serum naltrexone prior to dosing and at times 2, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 hours after naltrexone administration
Plasma Concentration (AUC 0-inf) | 48 hours
  Measurement of serum naltrexone prior to dosing and at times 2, 3, 4, 6, 8, 12, 16, 24, 30, 36 and 48 hours after naltrexone administration

SECONDARY OUTCOMES:
Adverse Events | Maximum of 18 days
  Will be reported from the start of the first session to follow-up visit
Vital Signs | 12 days
  Measured before and after naltrexone administration
12-lead electrocardiogram | 12 days
  Measured before and after naltrexone administration
Nasal Irritation Scoring | 5 days
  Will be reported from the start of the first session to follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Nora Chiang, PhD, Study Chair — National Institute on Drug Abuse (NIDA)
Locations (1):
- Vince and Associates Clinical Research, Inc., Overland Park, Kansas, United States